CLINICAL TRIAL: NCT00215046
Title: Vinblastine and Methotrexate in Children With Multivessel Pulmonary Vein Stenosis-A Phase II Study
Brief Title: Vinblastine and Methotrexate in Children With Pulmonary Vein Stenosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Mark Kieran/ Director, Neuro Oncology, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH 02-04-054 R
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Intraluminal Pulmonary Vein Stenosis
Keywords: vinblastine; methotrexate
MeSH Terms: interventions — Vinblastine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug (Experimental): no randomization, all patients receive experimental drugs
  Interventions: Drug: Vinblastine; Drug: Methotrexate

INTERVENTIONS:
Drug: Vinblastine — drug - dosage and frequency is based on size of patient and response to treatment.
  Other Names: antimicrotubule drug
Drug: Methotrexate — drug - dosage is based on size of patient and frequency and duration is based on response to treatment.
  Other Names: Trexall

SUMMARY:
To evaluate the efficacy of the chemotherapeutic agents vinblastine and methotrexate in the treatment of two groups of children with multivessel pulmonary vein stenosis. Group 1 will contain children with multivessel pulmonary vein stenosis who do not have structural heart disease, and Group 2 will consist of children with multivessel pulmonary vein stenosis and concomitant structural heart disease.

The primary outcome variable for efficacy is patient status one year after the start of treatment, where status is classified as either failure or success. Failure is defined as death or evidence of progressive obstruction at any time over the course of treatment as defined in the protocol. Success constitutes complete or partial response to treatment or stability of disease. Secondary outcome variables for efficacy are survival, time from diagnosis of pulmonary vein stenosis until failure, and change in patient classification on a scale measuring the severity of the obstructive disease.

1.2 To assess the safety of vinblastine and methotrexate in the treatment of multivessel pulmonary vein stenosis.

The primary outcome variable for safety is any occurrence of toxicity related to the administration of the chemotherapeutic agents over the treatment period.

DETAILED DESCRIPTION:
We sought to develop a regimen that might successfully suppress myofibroblastic proliferation in infants and children with progressive pulmonary vein stenosis. A number of factors need to be considered when proposing novel treatment options for patients with multivessel pulmonary vein stenosis. Specifically:

* Treatment should be directed against a specific target, in this case excessive proliferation of myofibroblasts.
* Treatment should have known activity against the target cell.
* Treatment should be well-tolerated in the patient group. In this case, agents with minimal hemodynamic side effects would be preferred.
* Treatment should not preclude patients from participation in other potentially effective therapies. Specifically, agents that do not cause significant myelosuppression would allow listing for transplantation.
* Treatment should not interfere with normal growth and development, and should have minimal if any risk for long-term toxicity or second tumors.

After considering these factors, we chose to administer two chemotherapeutic agents, vinblastine and methotrexate. Vinblastine and methotrexate have over 30 years of usage and are well-tolerated. The agents used are given in low-dose and do not usually cause nausea or vomiting, nor do they cause significant immunosuppression which, if present, could lead to a risk of infection and fever.

Desmoid tumors, also referred to as infantile fibromatosis, overlap with infantile myofibromatosis. A combination of standard agents that has been successfully used to treat desmoid tumors in infants is vinblastine and methotrexate (24). As opposed to cyclophosphamide-based regimens, this combination has the distinct advantages of few acute side effects and no known long-term toxicities, such as infertility or second malignancy. These agents have been used for over 30 years to treat infant and childhood malignancies. Over the last five years, methotrexate and vinblastine have been used to treat 9 children with recurrent desmoid tumor, a lesion similar although not identical to the abnormality present in patients with pulmonary vein stenosis. This regimen had minimal acute toxicity limited to mild to moderate nausea (which is easily controlled with anti-emetic therapy), minimal alopecia, mild hepatic inflammation, and mild myelosuppression. An addition advantage is that these drugs do not interfere with listing for lung transplantation, an important factor in the overall treatment options for this patient population. Instead of high-dose administration of chemotherapy (that catches only those cells in cycle at the time of administration), the low-dose chronic weekly administration continues to catch proliferating cells as they continually come into cycle. This may explain why the only other trial of chemotherapy (with high-dose cytoxan) was unsuccessful. Of the 9 children with desmoid lesions who received vinblastine and methotrexate therapy, four patients were treated for 18 months or longer. At the time of the last report, no patient had progressive disease during therapy. Two children had radiographically stable disease 1 and 2 years after treatment. Two children had stable disease for 1 and 2 years after treatment and then had disease progression. Thus, this drug combination is well-tolerated, has minimal side effects, and has demonstrated clinical activity against a closely related type of lesion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis can be based on clinical and radiographic grounds or at the time of biopsy or prior surgical procedures. The diagnosis must be consistent with multivessel pulmonary stenosis.
* There must be evidence of severe pulmonary vein stenosis in at least two pulmonary veins.
* Evidence of myofibroblast neo-proliferation, if biopsies were obtained.
* Staging must include a complete cardiovascular evaluation including echocardiogram, and EKG.
* Accepted organ function includes:

  * Creatinine < 1.5 x normal for age.
  * SGPT, Bilirubin < 1.5 x normal for age.
  * ANC ³ 1,500/mm3, Hemoglobin ³ 10g/dl, Platelets ³ 100,000/mm3
* Placement of a permanent central venous line. CVL access is necessary in all patients as vinblastine is a vesicant and will cause a tissue burn if infiltrated into the skin. Because a CVL may interfere with proper cardiac assessment in this patient population, the study physician will be made aware prior to the placement of a line.
* Patients may be listed for a lung transplant while enrolled on this study.
* All patients must have given written informed consent according to institutional guidelines.

Exclusion Criteria:

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2000-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable for efficacy is patient status one year after the start of treatment, where status is classified as either failure or success. Failure is defined as death or evidence of progressive obstruction at any time over the course of | 1 year
  Clinical status is assessed at one year for efficacy. Additionally, the toxicity are assessed at this time for the safety endpoint.

SECONDARY OUTCOMES:
Secondary outcome variables for efficacy are survival, time from diagnosis of pulmonary vein stenosis until failure, and change in patient classification on a scale measuring the severity of the obstructive disease. | 1 year
  Survival is evaluated one year after starting treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Kieran, MD,PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts